CLINICAL TRIAL: NCT01653457
Title: Efficacy of Memantine in the Treatment of Fibromyalgia: a Double-blind Randomized Trial
Brief Title: Randomised Controlled Trial of Memantine in Fibromyalgia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aragon Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC11-387
Record Dates: First submitted 2012-07-06; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Magnetic Resonance Spectroscopy; Memantine; electroencephalic cordance
MeSH Terms: conditions — Fibromyalgia | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Memantine (Active Comparator)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Patients randomised to this arm will receive memantine 20 mg daily. This dose will be reached following this schema:
  * 1st week: 5 mg daily
  * 2nd week: 10 mg daily
  * 3rd week: 15 mg daily
  * From 4th week up to 24th week: 20 mg daily
  Other Names: Ebixa
  Arms: Memantine
Drug: Placebo — Patients randomised to this group will receive film-coated placebo tablets (similar to drug tablets.
  Arms: Placebo

SUMMARY:
Fibromyalgia (FM) is a chronic rheumatic disease of high prevalence and great clinical impact. However, the treatment for FM has limited efficacy, with an effect size of about 0.5. Recent studies have found raised levels of glutamate in the insula, hippocampus and posterior cingulate cortex regions of the brain. This has led a number of authors to suggest the usefulness of glutamate blocking drugs in the treatment of FM.

Aims: To evaluate the efficacy of memantine in the treatment of pain and other symptoms of FM and to assess its efficacy in reducing brain glutamate levels in patients with FM. Material and methods: Randomized controlled trial, of six months duration (including a dose adjustment period of one month). 60 patients with FM will be recruited for inclusion in the study upon fulfillment of selection criteria, and they will be randomized in two groups: A) Treatment group (n=30), will receive 20 mg of memantine o.d ; B) Control group (n=30) will receive placebo. The main objective is to assess the efficacy of memantine in the treatment of pain (pain threshold, pain perception) and other symptoms in fibromyalgia (cognitive state, health status, state of anxiety and depression, quality of life and perceived improvement. Discussion: There is a need for the development of innovative and more effective alternatives for the treatment of FM. This clinical trial will determine whether memantine can be considered as an option in the treatment of FM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 65 years.
2. Ability to understand Spanish.
3. Diagnosis of fibromyalgia carried out by a rheumatologist according to the American College of rheumatology criteria (ACR1990).
4. Ability to read and understand the Patient Information Sheet
5. Signature of Informed Consent Form.

6 .In the case of women of childbearing age, commitment not to become pregnant during the entire duration of the study.

Exclusion Criteria:

1. Undergoing drug treatment for fibromyalgia. Patients undergoing treatment for fibromyalgia will stop treatment and perform a washout period of one week. During that week the patient may take, if necessary, analgesic such as paracetamol, ibuprofen and other NSAIDS to minimize the influence of medication on brain imaging.
2. Currently taking memantine or having taken memantine during the 2 months prior to recruitment.
3. Another Axis I psychiatric disorder using SCID-I that might hinder adherence to the protocol (e.g.: dementia, alcohol and/or substance abuse/dependence, schizophrenia, chronic delirium, acute depression).
4. Pregnancy or breast-feeding.
5. Hypersensitivity to the active ingredient, memantine, or to the excipients.
6. Medical conditions that require special precautions when administering memantine according to the summary of product characteristics:

   * Epilepsy.
   * Circumstances that may cause high urine pH owing to Proteus urinary infection, renal tubular acidosis or vegetarian diet, recent myocardial infarction, congestive heart disease and uncontrolled arterial hypertension.
7. Clinically significant and active evidence of liver or kidney disease, haematological, respiratory, endocrine or cardiovascular disease or disorders (patients with controlled diabetes and patients with controlled hypertension and complete or incomplete right bundle branch block can be included in the study).
8. Use of prescription drugs that may cause relevant drug interactions with memantine according to the summary of product characteristics: NMDAR antagonists (amantadine, ketamine, dextromethorphan), L-Dopa, dopamine agonists and cholinergic agonists.
9. Use of non-permitted concomitant medication during the week prior to the first evaluation visit or when the patient is expected to require treatment (with at least one of the drugs not permitted during the study): antidepressants (duloxetine, venlafaxine, mirtazapine, bupropion, SSRI, etc.), analgesics (pregabalin, gabapentin, opiates, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-10 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain threshold at month 1 | Month 1
  It will be measured by sphygmomanometry, a clinical test widely used and very efficient to identify patients with fibromyalgia.
Change from baseline in pain threshold at month 3 | Month 3
  It will be measured by sphygmomanometry, a clinical test widely used and very efficient to identify patients with fibromyalgia. Pain perception will be evaluated with the Pain Visual Analogue Scale (VAS pain). It is a horizontal line, 10 cm in length, anchored by word descriptors at each end (no pain and very severe pain)
Change from baseline in pain threshold at month 6 | Month 6
  It will be measured by sphygmomanometry, a clinical test widely used and very efficient to identify patients with fibromyalgia.
Change from baseline in pain perception at month 1 | Month 1
  Pain perception will be evaluated with the Pain Visual Analogue Scale (VAS pain). It is a horizontal line, 10 cm in length, anchored by word descriptors at each end (no pain and very severe pain)
Change from baseline in pain perception at month 3 | Month 3
  Pain perception will be evaluated with the Pain Visual Analogue Scale (VAS pain). It is a horizontal line, 10 cm in length, anchored by word descriptors at each end (no pain and very severe pain)
Change from baseline in pain perception at month 6 | Month 6
  Pain perception will be evaluated with the Pain Visual Analogue Scale (VAS pain). It is a horizontal line, 10 cm in length, anchored by word descriptors at each end (no pain and very severe pain)

SECONDARY OUTCOMES:
To assess improvement in cognitive state | Baseline, month 1, month 3 and month 6
  It will be measured by the Cognition Mini-Exam (MEC).In people under 65 years old, like the population in our study, the threshold that suggests a "probable case" is <27 points. The Spanish version of the questionnaire will be used.
  Cognitive state will also be measured by qEEG event-related desynchronization (ERD) at absolute power of upper alpha rhythms in the parieto-occipital region while cognitive tasks are performed.
To assess improvement in Health Status | Baseline, month 1, month 3 and month 6
  It will be evaluated with the Fibromyalgia Impact Questionnaire (FIQ). FIQ is a 10-Item self-questionnaire to measure the Health Status in patients with fibromyalgia. The Spanish version will be used.
To assess Anxiety and depression levels | Baseline, month 1, month 3 and month 6
  This will be evaluated with the Hospital Anxiety Depression Scale (HADS).Spanish version will be used.
To assess Quality of life | Baseline, month 1, month 3 and month 6
  It will be measured by the EuroQol 5D questionnaire. Spanish version will be used.
To assess Clinical Global Impression | Baseline, month 1, month 3 and month 6
  It will be evaluated with the Clinical Global Impression scale.
Glutamate levels in different brain regions (insula, hippocampus and posterior cingulate cortex). | Baseline, month 6
  This will be assessed with magnetic resonance spectroscopy (MRS) and by quantitative encephalography and electroencephalic cordance.

CONTACTS AND LOCATIONS:
Overall Officials: José Javier García Campayo, PhD, Principal Investigator — Miguel Servet University Hospital
Locations (1):
- Mental Health Unit, Primary Care Center "Torrero"., Zaragoza, Zaragoza, Spain

REFERENCES:
- [Background] Staud R, Vierck CJ, Robinson ME, Price DD. Effects of the N-methyl-D-aspartate receptor antagonist dextromethorphan on temporal summation of pain are similar in fibromyalgia patients and normal control subjects. J Pain. 2005 May;6(5):323-32. doi: 10.1016/j.jpain.2005.01.357. PMID 15890634
- [Background] Graven-Nielsen T, Kendall SA, Henriksson KG, Bengtsson M, Sorensen J, Johnson A, Gerdle B, Arendt-Nielsen L. Ketamine reduces muscle pain, temporal summation, and referred pain in fibromyalgia patients. Pain. 2000 Apr;85(3):483-491. doi: 10.1016/S0304-3959(99)00308-5. PMID 10781923
- [Background] Chen HS, Lipton SA. The chemical biology of clinically tolerated NMDA receptor antagonists. J Neurochem. 2006 Jun;97(6):1611-26. doi: 10.1111/j.1471-4159.2006.03991.x. PMID 16805772
- [Background] Tariot PN, Farlow MR, Grossberg GT, Graham SM, McDonald S, Gergel I; Memantine Study Group. Memantine treatment in patients with moderate to severe Alzheimer disease already receiving donepezil: a randomized controlled trial. JAMA. 2004 Jan 21;291(3):317-24. doi: 10.1001/jama.291.3.317. PMID 14734594
- [Background] Reisberg B, Doody R, Stoffler A, Schmitt F, Ferris S, Mobius HJ. A 24-week open-label extension study of memantine in moderate to severe Alzheimer disease. Arch Neurol. 2006 Jan;63(1):49-54. doi: 10.1001/archneur.63.1.49. PMID 16401736
- [Background] Nikolajsen L, Gottrup H, Kristensen AG, Jensen TS. Memantine (a N-methyl-D-aspartate receptor antagonist) in the treatment of neuropathic pain after amputation or surgery: a randomized, double-blinded, cross-over study. Anesth Analg. 2000 Oct;91(4):960-6. doi: 10.1097/00000539-200010000-00036. PMID 11004057
- [Background] Weinbroum AA, Rudick V, Paret G, Ben-Abraham R. The role of dextromethorphan in pain control. Can J Anaesth. 2000 Jun;47(6):585-96. doi: 10.1007/BF03018952. PMID 10875724
- [Background] Sinis N, Birbaumer N, Gustin S, Schwarz A, Bredanger S, Becker ST, Unertl K, Schaller HE, Haerle M. Memantine treatment of complex regional pain syndrome: a preliminary report of six cases. Clin J Pain. 2007 Mar-Apr;23(3):237-43. doi: 10.1097/AJP.0b013e31802f67a7. PMID 17314583
- [Background] Hackworth RJ, Tokarz KA, Fowler IM, Wallace SC, Stedje-Larsen ET. Profound pain reduction after induction of memantine treatment in two patients with severe phantom limb pain. Anesth Analg. 2008 Oct;107(4):1377-9. doi: 10.1213/ane.0b013e31817f90f1. PMID 18806054
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Gamero Ruiz F, Gabriel Sanchez R, Carbonell Abello J, Tornero Molina J, Sanchez-Magro I. [Pain in Spanish rheumatology outpatient offices: EPIDOR epidemiological study]. Rev Clin Esp. 2005 Apr;205(4):157-63. doi: 10.1157/13074161. Spanish. PMID 15860186
- [Background] Briley M. Drugs to treat fibromyalgia - the transatlantic difference. Curr Opin Investig Drugs. 2010 Jan;11(1):16-8. PMID 20047155
- [Background] Garcia-Campayo J, Magdalena J, Magallon R, Fernandez-Garcia E, Salas M, Andres E. A meta-analysis of the efficacy of fibromyalgia treatment according to level of care. Arthritis Res Ther. 2008;10(4):R81. doi: 10.1186/ar2455. Epub 2008 Jul 15. PMID 18627602
- [Background] Mountz JM, Bradley LA, Modell JG, Alexander RW, Triana-Alexander M, Aaron LA, Stewart KE, Alarcon GS, Mountz JD. Fibromyalgia in women. Abnormalities of regional cerebral blood flow in the thalamus and the caudate nucleus are associated with low pain threshold levels. Arthritis Rheum. 1995 Jul;38(7):926-38. doi: 10.1002/art.1780380708. PMID 7612042
- [Background] Kwiatek R, Barnden L, Tedman R, Jarrett R, Chew J, Rowe C, Pile K. Regional cerebral blood flow in fibromyalgia: single-photon-emission computed tomography evidence of reduction in the pontine tegmentum and thalami. Arthritis Rheum. 2000 Dec;43(12):2823-33. doi: 10.1002/1529-0131(200012)43:123.0.CO;2-E. PMID 11145042
- [Background] Garcia-Campayo J, Sanz-Carrillo C, Baringo T, Ceballos C. SPECT scan in somatization disorder patients: an exploratory study of eleven cases. Aust N Z J Psychiatry. 2001 Jun;35(3):359-63. doi: 10.1046/j.1440-1614.2001.00909.x. PMID 11437810
- [Background] Harris RE, Sundgren PC, Craig AD, Kirshenbaum E, Sen A, Napadow V, Clauw DJ. Elevated insular glutamate in fibromyalgia is associated with experimental pain. Arthritis Rheum. 2009 Oct;60(10):3146-52. doi: 10.1002/art.24849. PMID 19790053
- [Background] Choi DW, Koh JY, Peters S. Pharmacology of glutamate neurotoxicity in cortical cell culture: attenuation by NMDA antagonists. J Neurosci. 1988 Jan;8(1):185-96. doi: 10.1523/JNEUROSCI.08-01-00185.1988. PMID 2892896
- [Background] Leuchter AF, Cook IA, Lufkin RB, Dunkin J, Newton TF, Cummings JL, Mackey JK, Walter DO. Cordance: a new method for assessment of cerebral perfusion and metabolism using quantitative electroencephalography. Neuroimage. 1994 Jun;1(3):208-19. doi: 10.1006/nimg.1994.1006. PMID 9343572
- [Background] Leuchter AF, Uijtdehaage SH, Cook IA, O'Hara R, Mandelkern M. Relationship between brain electrical activity and cortical perfusion in normal subjects. Psychiatry Res. 1999 Apr 26;90(2):125-40. doi: 10.1016/s0925-4927(99)00006-2. PMID 10482384
- [Background] Cook IA, Leuchter AF, Morgan ML, Stubbeman W, Siegman B, Abrams M. Changes in prefrontal activity characterize clinical response in SSRI nonresponders: a pilot study. J Psychiatr Res. 2005 Sep;39(5):461-6. doi: 10.1016/j.jpsychires.2004.12.002. PMID 15992554
- [Background] Venneman S, Leuchter A, Bartzokis G, Beckson M, Simon SL, Schaefer M, Rawson R, Newton T, Cook IA, Uijtdehaage S, Ling W. Variation in neurophysiological function and evidence of quantitative electroencephalogram discordance: predicting cocaine-dependent treatment attrition. J Neuropsychiatry Clin Neurosci. 2006 Spring;18(2):208-16. doi: 10.1176/jnp.2006.18.2.208. PMID 16720798
- [Background] Hunter AM, Leuchter AF, Morgan ML, Cook IA. Changes in brain function (quantitative EEG cordance) during placebo lead-in and treatment outcomes in clinical trials for major depression. Am J Psychiatry. 2006 Aug;163(8):1426-32. doi: 10.1176/ajp.2006.163.8.1426. PMID 16877657
- [Background] Evans KC, Dougherty DD, Pollack MH, Rauch SL. Using neuroimaging to predict treatment response in mood and anxiety disorders. Ann Clin Psychiatry. 2006 Jan-Mar;18(1):33-42. doi: 10.1080/10401230500464661. PMID 16517451
- [Background] Bares M, Brunovsky M, Kopecek M, Stopkova P, Novak T, Kozeny J, Hoschl C. Changes in QEEG prefrontal cordance as a predictor of response to antidepressants in patients with treatment resistant depressive disorder: a pilot study. J Psychiatr Res. 2007 Apr-Jun;41(3-4):319-25. doi: 10.1016/j.jpsychires.2006.06.005. Epub 2006 Aug 4. PMID 16889798
- [Background] Bares M, Brunovsky M, Kopecek M, Novak T, Stopkova P, Kozeny J, Sos P, Krajca V, Hoschl C. Early reduction in prefrontal theta QEEG cordance value predicts response to venlafaxine treatment in patients with resistant depressive disorder. Eur Psychiatry. 2008 Aug;23(5):350-5. doi: 10.1016/j.eurpsy.2008.03.001. Epub 2008 May 2. PMID 18450430
- [Background] Vargas A, Vargas A, Hernandez-Paz R, Sanchez-Huerta JM, Romero-Ramirez R, Amezcua-Guerra L, Kooh M, Nava A, Pineda C, Rodriguez-Leal G, Martinez-Lavin M. Sphygmomanometry-evoked allodynia--a simple bedside test indicative of fibromyalgia: a multicenter developmental study. J Clin Rheumatol. 2006 Dec;12(6):272-4. doi: 10.1097/01.rhu.0000249770.86652.3b. PMID 17149055
- [Background] Sriwatanakul K, Kelvie W, Lasagna L, Calimlim JF, Weis OF, Mehta G. Studies with different types of visual analog scales for measurement of pain. Clin Pharmacol Ther. 1983 Aug;34(2):234-9. doi: 10.1038/clpt.1983.159. PMID 6872418
- [Background] Lobo A, Saz P, Marcos G, Dia JL, de la Camara C, Ventura T, Morales Asin F, Fernando Pascual L, Montanes JA, Aznar S. [Revalidation and standardization of the cognition mini-exam (first Spanish version of the Mini-Mental Status Examination) in the general geriatric population]. Med Clin (Barc). 1999 Jun 5;112(20):767-74. Spanish. PMID 10422057
- [Background] Klimesch W, Doppelmayr M, Hanslmayr S. Upper alpha ERD and absolute power: their meaning for memory performance. Prog Brain Res. 2006;159:151-65. doi: 10.1016/S0079-6123(06)59010-7. PMID 17071229
- [Background] Rivera J, Gonzalez T. The Fibromyalgia Impact Questionnaire: a validated Spanish version to assess the health status in women with fibromyalgia. Clin Exp Rheumatol. 2004 Sep-Oct;22(5):554-60. PMID 15485007